CLINICAL TRIAL: NCT06120062
Title: The Effect of Swaddling and Inhaling Breast Milk Odour on the Pain and Comfort During the Placement of Peripheral Intravenous Catheter in Term Infants
Brief Title: Effect of Swaddling and Inhaling Breast Milk Odour on the Pain and Comfort
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Ayla Gündoğdu Karakaya, Doctor of Pediatric Nursing, Zonguldak Bulent Ecevit University
Other Study IDs: 3272493AGK
Record Dates: First submitted 2023-02-19; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Infant, Newborn; Pain Perception
Keywords: newborn; pain; comfort; nurse; Non-pharmacological Method
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1st experimental group: swaddled
  Interventions: Other: swaddled
- 2nd experimental group: inhale the mother's breast milk odour
  Interventions: Other: mother's breast milk odor
- 3rd experimental group: both swaddled and made to inhale the mother's breast milk odour
  Interventions: Other: both swaddled and made to inhale mother's breast milk odor
- the control group: no procedure
  Interventions: Other: No procedure

INTERVENTIONS:
Other: swaddled — the 1st experimental group were swaddled
  Groups: 1st experimental group
Other: mother's breast milk odor — the 2nd experimental group were made to inhale mother's breast milk odor
  Groups: 2nd experimental group
Other: both swaddled and made to inhale mother's breast milk odor — the 3rd experimental group were both swaddled and made to inhale mother's breast milk odor
  Groups: 3rd experimental group
Other: No procedure — No procedure was applied to the infants in the control group.
  Groups: the control group

SUMMARY:
This randomized controlled experimental study was conducted to determine the effect of swaddling and inhaling mother's breast milk odour on the pain and comfort during the placement of peripheral intravenous catheter in term infants.The population of the study consisted of term infants hospitalized in the neonatal intensive care unit of Karadeniz Ereğli State Hospital between 1st October 2020 and 1st October 2021. According to the G-Power analysis, the sample size was calculated as 120 and term infants were equally assigned to three experimental groups and a control group, each of which consisted of 30 infants. During the placement of peripheral intravenous catheter, the infants in the 1st experimental group were swaddled, the infants in the 2ndexperimentalgroup were made to inhale the mother's breast milk odour, the infants in the 3rd experimental group were both swaddled and made to inhale the mother's breast milk odour and no procedure was applied to the infants in the control group. The pain and comfort levels of infants in the experimental and control groups were assessed before, during and after the placement of peripheral intravenous catheter. "Infant Descriptive Information Form", "Neonatal Infant Pain Scale (NIPS)" and "Neonatal Comfort Behaviour Scale (NCBS) were used to collect data.

DETAILED DESCRIPTION:
The effect of Swaddling and Inhaling Breast Milk Odour on the Pain and Comfort During the Placement of Peripheral Intravenous Catheter in Term Infants.

This randomized controlled experimental study was conducted to determine the effect of swaddling and inhaling mother's breast milk odour on the pain and comfort during the placement of peripheral intravenous catheter in term infants.

The population of the study consisted of term infants hospitalized in the neonatal intensive care unit of Karadeniz Ereğli State Hospital between 1st October 2020 and 1st October 2021. According to the G-Power analysis, the sample size was calculated as 120 and term infants were equallyassigned to three experimental groups and a control group, each of which consisted of 30 infants. During the placement of peripheral intravenous catheter, the infants in the 1st experimental group were swaddled, the infants in the 2ndexperimentalgroup were made to inhale the mother's breast milk odour, the infants in the 3rd experimentalgroup were both swaddled and made to inhale the mother's breast milkodour and no procedure was applied to the infants in the control group. The pain and comfort levels of infants in the experimental and control groups were assessed before, during and after the placement of peripheral intravenous catheter."Infant Descriptive Information Form", "Neonatal Infant Pain Scale" and "Neonatal Comfort Behaviour Scale were used to collect data.

ELIGIBILITY:
Sample selection criteria of the study

* Being a term infant (born at 37-41 weeks of gestation)
* Being currently hospitalized in the neonatal intensive care unit
* Not having a previous insertion of peripheral intravenous catheter
* Having the insertion of peripheral intravenous catheter for the first time
* Having no invasive procedures before (insertion of peripheral intravenous catheter, urethral Foley catheterisation, nasogastric tube insertion, etc.)
* Having no analgesic before the procedure

Exclusion criteria of the study

* Refusing to participate in the research
* Having been given analgesics
* Inability to open the vascular access in one go

Ages: 1 Day to 27 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 120 and term infants were equallyassigned to three experimental groups and a control group, each of which consisted of 30 infants
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
the effect of swaddling the pain and comfort during the placement of peripheral intravenous catheter | 20 minutes
  Infants in the 1st experimental group (Swaddling) were swaddled when they were laid under a radiant heater for the insertion of peripheral intravenous catheter. The Neonatal Infant Pain Scale (NIPS) and the Newborn Comfort Behavior Scale were evaluated by the researcher before and during the procedure, and 5 minutes after they were taken into the incubator.

SECONDARY OUTCOMES:
the effect of inhaling mother's breast milk odour on the pain and comfort during the placement of peripheral intravenous catheter | 20 minutes
  Infants in the 2nd experimental group (Inhaling mother's breast milk odor) were made to inhale their mothers' breast milk odor when they were laid under a radiant heater for the insertion of peripheral intravenous catheter. The Neonatal Infant Pain Scale (NIPS) and the Newborn Comfort Behavior Scale were evaluated by the researcher before and during the procedure, and 5 minutes after they were taken into the incubator.

OTHER OUTCOMES:
the effect of both swaddled and made to inhale mother's breast milk odor. | 20 minutes
  Infants in the 3rd experimental group (Swaddling and inhaling mother's breast milk odor) were both swaddled and made to inhale their mothers' breast milk odor when they were laid under a radiant heater for the insertion of peripheral intravenous catheter. The Neonatal Infant Pain Scale (NIPS) and the Newborn Comfort Behavior Scale were evaluated by the researcher before and during the procedure, and 5 minutes after they were taken into the incubator.

CONTACTS AND LOCATIONS:
Overall Officials: ayla gündoğdu karakaya, Study Director — zonguldak beun
Locations (1):
- zonguldak BEU, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rad ZA, Aziznejadroshan P, Amiri AS, Ahangar HG, Valizadehchari Z. The effect of inhaling mother's breast milk odor on the behavioral responses to pain caused by hepatitis B vaccine in preterm infants: a randomized clinical trial. BMC Pediatr. 2021 Feb 1;21(1):61. doi: 10.1186/s12887-021-02519-0. PMID 33522927
- [Result] Lan HY, Yang L, Lin CH, Hsieh KH, Chang YC, Yin T. Breastmilk as a Multisensory Intervention for Relieving Pain during Newborn Screening Procedures: A Randomized Control Trial. Int J Environ Res Public Health. 2021 Dec 10;18(24):13023. doi: 10.3390/ijerph182413023. PMID 34948633
- [Result] Yilmaz D, Inal S. Effects of three different methods used during heel lance procedures on pain level in term neonates. Jpn J Nurs Sci. 2020 Oct;17(4):e12338. doi: 10.1111/jjns.12338. Epub 2020 Apr 2. PMID 32239753
- See also: national thesis center — http://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp